CLINICAL TRIAL: NCT04906954
Title: Effects of Combining a Neuromuscular Electrical Stimulation Intervention With Nutritional Support in Deconditioned Patients With Advanced Gastrointestinal Cancer - DIG'ELECTROSTIM-01
Brief Title: Combined Neuromuscular Electrical Stimulation and Nutritional Support for Advanced Gastrointestinal Cancer Patients.
Acronym: DIGELECTROSTIM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not initiated due to logistical challenges, and the contract for the acquisition of the equipment-comprising relatively high-cost machinery-was never finalized.
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DIG' ELECTROSTIM-01-G-097
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Cancer Digestive
Keywords: electrostimulation
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase II
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neuromuscular electrical stimulation (NMES) (Other): 30 NMES sessions will be performed by patients for 30 min, for a period of 8 weeks, according to a standardized protocol.
  The number of sessions per week will be gradually increased to reach 5 sessions/week at week 4.
  Interventions: Other: NMES

INTERVENTIONS:
Other: NMES — Standardized strength program (75 Hz frequency, 40 cycles). The stimulation intensity will be increased up to the highest tolerated level in order to evoke strong muscle contractions.

SUMMARY:
Dig' Electrostim-01 is phase II, single center (step 1) and multicentre (step 2), single-arm study to evaluate an 8-week NMES intervention combined with nutritional support in addition to usual patient care

DETAILED DESCRIPTION:
Sarcopenia and cachexia are observed in more than 50% of patients with gastrointestinal (GI) cancer.

Both negatively affect patient survival and health-related quality of life (HRQoL) due to decreased tolerance to anticancer treatments and increased susceptibility to infections and other complications. Therefore, sarcopenia and cachexia represent a major clinical issue in this setting. A multimodal therapeutic approach to the sarcopenia and cachexia management is recommended, including nutritional support and exercise with personalized oncology care and family-centered education.

Neuromuscular electrical stimulation (NMES) generates muscle contractions using portable devices connected to surface electrodes.

NMES is safe, does not require the active cooperation of the patient and can be self-administered at home, thereby providing an acceptable physical therapy for patients with advanced cancer and an altered Eastern Cooperative Oncology Group performance status (ECOG PS) and/or a high-symptom burden, for whom attendance to hospital-based exercise training is difficult.

In this study, we hypothesize that NMES is a safe and effective physical-therapy strategy to improve HRQoL and to reduce cancer-induced sarcopenia in patients with metastatic GI cancer and altered ECOG PS (ECOG PS of 2).

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent,
2. Age ≥ 18 years,
3. Mini Nutritional Assessment (MNA) and geriatric 8 (G8) health status screening tools for patients ≥ 70 years and oncogeriatric evaluation if G8 ≤ 14,
4. First-line chemotherapy for advanced disease,
5. Histologically confirmed colorectal, pancreatic, esophageal, or gastric cancer (adenocarcinoma or squamous cell carcinoma),
6. Metastatic disease not amenable to surgery, radiation, or combined modality therapy with curative intent (previous resection of primary tumor allowed),
7. Patients able to receive chemotherapy,
8. Eastern Cooperative Oncology Group performance status of 2,
9. Life expectancy ≥ 3 months,
10. Registration in a National Health Care System (Protection Universelle Maladie [PUMa] included).

Exclusion Criteria:

1. Neuroendocrine histology or primary tumor other than esophageal, gastric, pancreatic, biliary, or colorectal cancer,
2. Any medical (including psychiatric, musculoskeletal, or neurological) condition contra-indicating exercise practice,
3. Ulcerative skin lesions over the quadriceps muscle,
4. Participation to another physical activity program (exercise or NMES),
5. Pacemaker-depended patients,
6. Albuminemia < 25 g/L,
7. Pregnancy or breastfeeding,
8. Protected adults (individuals under guardianship by court order or tutelage). Note: participation to another concomitant clinical trial (except for trials evaluating exercise or NMES programs) is allowed, but the patient must inform about it and get an authorization from the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Step 1 : Number of patients who completed the neuromuscular electrical stimulation (NMES) program | At 6 months
  Step 1: Feasibility study will be performed on the first 10 patients. The NMES adherence will be satisfactory if the patient achieves ≥ 40% of planned sessions (12 in total). The NMES will be considered feasible if ≥ 70% of the first 10 patients included achieve this goal.
Step 2 : Number of patients with improvement of 10 points between baseline and week 8, assessed using the EORTC QLQ-C30 physical functioning scale | Up to 24 months
  At baseline, at week 8

SECONDARY OUTCOMES:
Time between inclusion and the observation of the first deterioration of at least 10 points as compared to the baseline score | Up to 24 months
  Every 2 moths until 12 months after inclusion
Progression-free survival (PFS) | Up to 24 months
  PFS defined as the time between inclusion and tumor progression (according to RECIST v1.1) or death (all causes), whichever occurs first
Overall Survival (OS) | Up to 24 months
  OS defined as the time between inclusion and death (from all causes)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy NEUZILLET, MD, Principal Investigator — Institut Curie Site Saint Cloud
Locations (1):
- Insitut Curie, Saint-Cloud, France

IPD SHARING:
Plan to Share IPD: No